CLINICAL TRIAL: NCT04948268
Title: Digital Mental Health Service for Non-Treatment Seeking Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Professor, Northwestern University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R34MH124960 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-07-01 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety; Suicidal Ideation
Keywords: Text messaging; Depression; Anxiety; Telemedicine; Digital Mental Health; mobile health (mHealth); Mobile phone; Technology assisted; Smartphone; Cell phone; Coach
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: This study uses a sequential multiple assignment randomized trial (SMART) design. The first level of randomization is to one of the three treatment conditions: self-guided non-personalized intervention, self-guided adaptive intervention, or active control. The second level of randomization occurs during the first two weeks of intervention. Participants who meet criteria for disengagement from either the non-personalized or adaptive intervention are then randomized to receive coaching or continue as self-guided. This will provide the investigators with preliminary information on the need for and value of coaching. Participants will receive the assigned intervention from baseline to week 8, followed by an 8 week follow-up period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Adaptive digital mental health intervention without coaching (Experimental): The adaptive intervention will consist of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Psychoeducational content will be delivered via a URL in an SMS message. Machine learning will be used to tailor messages and timing to meet participant preferences.
  Interventions: Behavioral: Adaptive messaging intervention
- Non-personalized digital Mental Health intervention without coaching (Experimental): The non-personalized intervention will consist of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Messages and content will not be tailored based on participants profile or usage.
  Interventions: Behavioral: Non-personalized messaging intervention
- Adaptive digital mental health intervention with coaching (Experimental): The adaptive intervention will consist of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Psychoeducational content will be delivered via a URL in an SMS message. Machine learning will be used to tailor messages and timing to meet participant preferences. Coaching will be provided to support engagement and intervention use via medium of participants choice (texts, calls, or emails).
  Interventions: Behavioral: Adaptive messaging intervention; Behavioral: Coaching
- Non-personalized digital Mental Health intervention with coaching (Experimental): The non-personalized intervention will consist of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Messages and content will not be tailored based on participants profile or usage. Coaching will be provided to support engagement and intervention use via medium of participants choice (texts, calls, or emails).
  Interventions: Behavioral: Non-personalized messaging intervention; Behavioral: Coaching
- Active control (Active Comparator): The active control condition will provide brief text messages that include a URL link to psychoeducational content, but will not include the interactive messaging component described in experimental arms.
  Interventions: Behavioral: Psychoeducational links

INTERVENTIONS:
Behavioral: Adaptive messaging intervention — Psychological content and messages delivered regularly over an 8-week period via interactive SMS messages. Content and messages will be tailored using machine learning.
  Arms: Adaptive digital mental health intervention with coaching; Adaptive digital mental health intervention without coaching
Behavioral: Non-personalized messaging intervention — Psychological content and messages delivered regularly over an 8-week period via interactive SMS messages. Psychological content will center on a single psychological strategy each week. There will not be any tailoring of messaging and content based on group or individual level data.
  Arms: Non-personalized digital Mental Health intervention with coaching; Non-personalized digital Mental Health intervention without coaching
Behavioral: Coaching — Human coaching to support intervention use and engagement via telephone calls, text or email
  Arms: Adaptive digital mental health intervention with coaching; Non-personalized digital Mental Health intervention with coaching
Behavioral: Psychoeducational links — SMS messages with URLs containing brief psychoeducational information.
  Arms: Active control

SUMMARY:
This is a feasibility trial of a personalized 8-week text messaging intervention aimed at young adults (ages 18-25) with depression and anxiety who are not interested in -- or experience barriers to -- receiving traditional face-to-face psychological treatments.

The trial will consist of a pilot test of (1) an 8-week adaptive (personalized) messaging intervention relative to (2) a non-personalized digital mental health intervention, or (3) an active control which will send weekly psychoeducation information by way of Uniform Resource Locators (URLs). The adaptive intervention will uses machine learning to tailor Short Message Service (SMS) messages to an individual's needs and preferences, and URL links to provide access to psychoeducational content to contextualize messages, when the length of that content exceeds the limitations of messages.

The primary goals of the project are to conduct a feasibility trial using a sequential multiple assignment randomized treatment (SMART) design, which will evaluate (a) the effectiveness of an adaptive, personalized messaging intervention in reducing engagement relative to a non-personalized version; and (b) whether human coaching results in greater symptom reduction and engagement, relative an unguided implementation.

DETAILED DESCRIPTION:
The primary purpose of this trial is to test the feasibility of conducting a randomized controlled trial of digital mental health intervention (DMHI) for non-treatment seeking young adults with symptoms of depression or anxiety, comparing an 8-week adaptive (personalized) messaging intervention, an 8-week non-personalized digital mental health intervention, or an active control which will deliver psychoeducational content via clickable URLs. The adaptive intervention will be powered by reinforcement learning to deliver tailored SMS messages based on user profiles and the ways in which a user interacts with the intervention system, along with links to longer psychoeducational content. The non-personalized intervention arm will not personalize the messages, but will still be an active treatment. This study will examine the adaptive intervention's ability to engage users and effectiveness in decreasing psychological distress relative to a non-personalized intervention. Participants who become disengaged (5 continuous days of not clicking on content URL links, responding to messages, or message ratings) from the adaptive or static intervention arms at any point in the first two weeks of treatment will be randomized to receive low-intensity human coaching or continue without coaching for the remainder of the intervention period.

Recruitment will take place via Mental Health America's (MHA) website. MHA is a large mental health advocacy organization that hosts online screeners and has large number of visitors the majority of whom meet clinical cutoffs for depressive or anxiety disorder symptoms. This study will enroll individuals who have completed a depression or anxiety disorder screener on MHA's website, and meet clinical cut-offs on the Patient Health Questionnaire - 9 (PHQ-9) or Generalized Anxiety Disorder - 7 (GAD-7).

Initial randomization will be generated in permuted blocks of 5 using a computer program. To prevent allocation bias, randomization will be conducted by the biostatistician, who will not inform the study team of the treatment arms until the baseline assessment has been completed and the patient has been enrolled. Second randomization of disengaged participants will occur as disengagement is detected during the first two weeks. Half (50%) of disengaged individuals will be randomized to receive additional human coaching throughout the remainder of the study while remaining in either the adaptive or non-personalized treatment arms. The disengaged participants not randomized to receive additional human coaching will continue to receive either the non-personalized or adaptive automated treatment the participants were randomized to initially.

Coaching will consist of providing users with support and accountability via positive reinforcement, goal and expectation setting, and monitoring. Coaching outreach will focus on adherence to the treatment but will not provide treatment advice. Coaches will provide a brief (15-minute phone call or equivalent depending on the medium) engagement session over the phone, SMS, or email, depending user preference. Thereafter, coaches will check in with participants via messaging, phone call, or email, twice per week and respond to patient texts.

Participants will be assessed using self-report measures at baseline, weeks 4, 8, 12, and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 25 *The age to provide consent in Nebraska is 19. Individuals recruited from the state of Nebraska must be 19 or older.
2. A positive screen on an MHA screen for depression (Patient Health Questionnaire - 9 [PHQ-9]) or anxiety (Generalized Anxiety Disorder - 7 [GAD-7]);
3. Resident of the United States.
4. Owns a smartphone

Exclusion Criteria:

1. Current treatment with psychotherapy or psychiatric medication management;
2. Seeking or plans to seek traditional mental health treatment (psychotherapy or psychiatric medication management) in next 8 weeks;
3. Serious mental illness for which intervention would be contraindicated (e.g., psychotic disorder, manic episode, etc.)
4. Severe suicidality (i.e., experiencing suicidal ideation with a plan and intent to act);
5. English insufficient to engage in design activities.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through and managed by the National Institute of Mental Health (NIMH) Data Archive (NDA). De-identified human subjects data, harmonized to a common standard, are available to qualified researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available after publication of the primary outcome papers.
Access Criteria: The NIMH Data Archive is managed by the NIMH. Access criteria are determined by the NIMH.
URL: https://nda.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Mental Health America (MHA) screening website. Website visitors who completed a depression or anxiety screening form and obtained a score of 10 or higher on either screener were eligible to see an advertisement for our study that contained a link to an informational page and eligibility screening form. Those meeting eligibility criteria were given an option of providing informed consent.
Pre-assignment Details: Prior to random assignment, participants who provided affirmative informed consent were required to have completed baseline assessments, confirm their ability to receive text messages as part of the intervention, and complete required payment forms.
Groups:
- Adaptive Digital Mental Health Intervention: The adaptive intervention will consist of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Psychoeducational content will be delivered via a URL in an SMS message. Machine learning will be used to tailor messages and timing to meet participant preferences.
- Non-personalized Digital Mental Health Intervention: The non-personalized intervention will consist of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Messages and content will not be tailored based on participants profile or usage.
Period: First Randomization
Arm/Group | Adaptive Digital Mental Health Intervention | Non-personalized Digital Mental Health Intervention | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Started | 40 | 40 | 0 | 0 | 40
Completed | 40 | 40 | 0 | 0 | 40
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Randomization
Arm/Group | Adaptive Digital Mental Health Intervention | Non-personalized Digital Mental Health Intervention | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Started | 34 | 30 | 6 | 10 | 40
Completed | 34 | 29 | 6 | 10 | 40
Not Completed | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Non-treatment seeking young adult Mental Health America website visitors
Groups:
- Total: Total of all reporting groups
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Active Control | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Grouping by initial treatment arm assignment
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 6 | 6 | 2 | 14
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 8 | 4 | 12
    White | 25 | 21 | 28 | 74
    More than one race | 5 | 4 | 5 | 14
    Unknown or Not Reported | 3 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Grouping by initial treatment arm assignment
  Participants
    Hispanic or Latino | 11 | 3 | 4 | 18
    Not Hispanic or Latino | 29 | 37 | 35 | 101
    Unknown or Not Reported | 0 | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants] — Population: Grouping by initial treatment arm assignment
  Participants
    <=18 years | 0 | 4 | 4 | 8
    Between 18 and 65 years | 40 | 36 | 36 | 112
    >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Grouping by initial treatment arm assignment
  Participants
    Participants Analyzed: Male | 7 | 9 | 6 | 22
    Participants Analyzed: Female | 28 | 30 | 31 | 89
    Participants Analyzed: Non-binary | 5 | 1 | 2 | 8
    Participants Analyzed: Self-describe | 0 | 0 | 1 | 1
Psychological Distress (Kessler 10/K10 Score) [Mean (Standard Deviation); unit: Score] — Population: Grouping by initial treatment arm assignment
  Score | 33.5 (6.77) | 31.125 (6.35) | 32.85 (6.88) | 32.49 (6.69)

OUTCOME MEASURES:

1. Primary Outcome: Kessler Psychological Distress Scale
Description: 10-item self-report measure of transdiagnostic distress, used as outcome measure across diagnostic categories. Higher scores mean greater distress. Minimum score: 10; maximum score: 50
Time Frame: 16 weeks
Population: Numbers are lower than participants assigned to groups due to loss to follow-up or incomplete data. Results are grouped per-arm and includes data from all participants with available data.
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Adaptive Digital Mental Health Intervention With Coaching: The adaptive intervention consists of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Psychoeducational content is delivered via a URL in an SMS message. Machine learning is be used to tailor messages and timing to meet participant preferences. Coaching is be provided to support engagement and intervention use via medium of participants choice (texts, calls, or emails).
- Non-personalized Digital Mental Health Intervention With Coaching: The non-personalized intervention consists of SMS messages, symptom tracking, and psychological content that centers on evidence-based psychological strategies. Messages and content are nottailored based on participants profile or usage. Coaching is provided to support engagement and intervention use via medium of participants choice (texts, calls, or emails).
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 29 | 24 | 6 | 9 | 31
Score | 23.52 (5.47) | 23.54 (7.84) | 24.50 (8.02) | 23.78 (5.43) | 26.58 (8.32)

2. Primary Outcome: Engagement Length
Description: Last message/content rating or click on content URL link received from participant. This measure can include select individuals who exceed 56 days of interaction due to user's ability to temporarily pause receipt of messages, resulting in messages extending beyond 8 weeks (56 days).
Time Frame: 62 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 34 | 30 | 6 | 10 | 40
Days | 51.4 (89.4) | 54.2 (7.27) | 36.2 (17.3) | 56.2 (29.7) | 50.1 (58.2)

3. Secondary Outcome: Patient Health Questionnaire-9
Description: 10-item self-report measure assessing depression symptom severity. Higher scores mean greater symptom severity. Minimum score: 0; maximum score: 27
Time Frame: 16 weeks
Population: Differences in numbers from those assigned due to loss to follow-up or individuals with incomplete data. Results are grouped per arm and include data from all participants with available data.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 29 | 24 | 6 | 8 | 30
Score | 9.59 (4.79) | 8.79 (5.15) | 9.83 (9.28) | 9.50 (5.15) | 11.77 (7.21)

4. Secondary Outcome: Generalized Anxiety Disorder-7
Description: 8-item self-report measure assessing generalized anxiety disorder symptom severity Higher scores mean greater symptom severity. Minimum score: 0; maximum score: 21
Time Frame: 16 weeks
Population: Numbers are lower than participants assigned to groups due to loss to follow-up or incomplete data. Results are grouped per arm and include data from all participants with available data.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 29 | 24 | 6 | 8 | 30
Score | 7.93 (3.83) | 7.54 (5.80) | 4.67 (4.27) | 7.37 (4.10) | 9.47 (5.85)

5. Other Pre Specified Outcome: Depression Symptom Inventory - Suicidality Subscale
Description: 4-item self-report questionnaire assessing the frequency and intensity of suicidal thoughts over previous two weeks.
  Higher scores signal greater frequency and severity of suicidal thoughts. Minimum score: 0; maximum score: 12
Time Frame: 16 weeks
Population: Numbers are lower than participants assigned to groups due to loss to follow-up or incomplete data. Results are grouped per arm and thus include data from all participants with available data.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 29 | 24 | 6 | 8 | 30
Score | 0.34 (1.17) | 0.17 (0.64) | 1.00 (1.26) | 0.75 (1.39) | 1.13 (1.94)

6. Other Pre Specified Outcome: Cognitive Behavioral Response to Stress Scale
Description: 9-item self-report measure of behavioral and cognitive coping related skills. Higher scores indicate greater adaptive cognitive and behavioral skills use.
  Two domains: Frequency of use and usefulness. For each domain, there is a subscale of cognitive (4 items) or behavioral (5 items) coping skills. Frequency rated 0-6 with higher scores being more frequent use. Usefulness is rated 0-6 with higher scores being more useful.
  Cognitive skill frequency range: 0-24 Cognitive skill usefulness range: 0-24 Behavioral skill frequency range: 0-35 Behavioral skill usefulness range: 0-35
Time Frame: 16 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 29 | 25 | 6 | 8 | 30
Score
  Cognitive Skill Frequency | 12.76 (4.13) | 12.37 (4.99) | 11.00 (6.63) | 8.75 (9.13) | 12.40 (4.38)
  Cognitive Skill Usefulness: number analyzed (Participants) | 25 | 25 | 5 | 4 | 25
  Cognitive Skill Usefulness | 11.04 (4.89) | 13.90 (5.52) | 11.60 (6.43) | 14.50 (7.51) | 12.52 (4.55)
  Behavioral Skill Frequency: number analyzed (Participants) | 29 | 24 | 6 | 8 | 30
  Behavioral Skill Frequency | 15.21 (4.77) | 16.42 (5.50) | 13.17 (5.27) | 10.62 (8.85) | 14.27 (4.29)
  Behavioral Skill Usefulness: number analyzed (Participants) | 22 | 17 | 4 | 4 | 20
  Behavioral Skill Usefulness | 18.27 (5.02) | 21.29 (5.20) | 17.00 (5.89) | 21.00 (3.74) | 18.30 (4.67)

7. Other Pre Specified Outcome: Objective Engagement Markers: Percent of Messages Responded to
Description: Number of messages responded to during the active messaging/intervention period.
Time Frame: 62 days
Population: Results are per arm and thus includes data from all participants with available data. This measure can include select individuals who exceed 56 days of interaction due to user's ability to temporarily pause receipt of messages, resulting in messages extending beyond 8 weeks (56 days). Because Active Control is not an interactive medium that contained messages to which participants could respond, there are no participants listed in the active control group.
Measure: Mean (Standard Deviation); unit: Percent of messages responded to
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 34 | 30 | 6 | 10 | 0
Percent of messages responded to | 53.7 (20.6) | 60.2 (25.2) | 18.7 (12.8) | 32.5 (18.6) |

8. Other Pre Specified Outcome: Objective Engagement Markers: Link Clicks
Description: Number of URL clicks during the study.
Time Frame: 62 days
Population: Results are grouped per arm. Means and standard deviations include only individuals with >0 link clicks. This measure can include select individuals who clicked on links beyond 56 days of interaction due to user's ability to temporarily pause receipt of messages.
Measure: Mean (Standard Deviation); unit: Number of link clicks per person
Arm/Group | Adaptive Digital Mental Health Intervention | Non-personalized Digital Mental Health Intervention | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
Number analyzed (Participants) | 27 | 26 | 4 | 6 | 34
Number of link clicks per person | 9.7 (20) | 9 (7.48) | 18 (22.6) | 4.83 (3.92) | 17.3 (12)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 16 weeks
Description: Results are grouped by initial treatment assignment (adaptive or non-personalized digital mental health intervention or control) as the primary focus of this feasibility trial was feasibility of primary treatment randomization and thus includes data from all participants.
Arm/Group | Adaptive Digital Mental Health Intervention Without Coaching | Non-personalized Digital Mental Health Intervention Without Coaching | Adaptive Digital Mental Health Intervention With Coaching | Non-personalized Digital Mental Health Intervention With Coaching | Active Control
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/30 | 0/6 | 0/10 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30 | 0/6 | 0/10 | 0/40
Other Adverse Events (participants affected / at risk) | 0/34 | 0/30 | 0/6 | 0/10 | 0/40

LIMITATIONS AND CAVEATS:
Loss to follow-up and missing data affect the interpretability of data from this trial (as all trials). Additionally, this trial was powered for feasibility not for efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04948268/Prot_000.pdf
  • Statistical Analysis Plan (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT04948268/SAP_001.pdf